CLINICAL TRIAL: NCT02013336
Title: Phase 1 Dose-escalating Study of MM-398 (Irinotecan Sucrosofate Liposome Injection) Plus Intravenous Cyclophosphamide in Recurrent or Refractory Pediatric Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Plains Oncology Consortium (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPOC-2012-001
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Recurrent or Refractory Solid Tumors; Ewing Sarcoma; Rhabdomyosarcoma; Neuroblastoma; Osteosarcoma
Keywords: pediatric; MM-398; cyclophosphamide; irinotecan
MeSH Terms: conditions — Recurrence; Sarcoma, Ewing; Rhabdomyosarcoma; Neuroblastoma; Osteosarcoma | interventions — irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MM-398 + cyclophosphamide (Experimental): MM-398+cyclophosphamide
  Interventions: Drug: MM-398 (Irinotecan Sucrosofate Liposome Injection) plus cyclophosphamide

INTERVENTIONS:
Drug: MM-398 (Irinotecan Sucrosofate Liposome Injection) plus cyclophosphamide — chemotherapy

SUMMARY:
This is a Phase 1 study of the combination of two drugs: MM-398 and Cyclophosphamide. The goal is to find the highest dose of MM-398 that can be given safely when it is used together with the chemotherapy drug Cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed Ewing sarcoma, rhabdomyosarcoma, neuroblastoma, or osteosarcoma
* Disease progression after prior therapy in locally advanced or metastatic setting
* Measurable or evaluable disease based on the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria
* Age 12 months to <21 years
* Adequate bone marrow reserves, hepatic function, and renal function
* Recovered from effects of any prior surgery or cancer therapy
* Patients 18 years or older will provide written consent. A parent or legal guardian of a patient <18 years of age will provide informed consent and patients 11 to 18 years of age will provide written assent or as per participating institutional policy.

Exclusion Criteria:

* Clinically significant gastrointestinal disorders
* NYHA Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure
* Active infection or unexplained fever
* Known hypersensitivity to any of the components of MM-398 or other liposomal products
* Recent Investigational therapy
* Pregnant or breast feeding; females of child-bearing potential must test negative for pregnancy at the time of enrollment

Ages: 12 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated Dose (MTD) of MM-398 in combination with intravenous cyclophosphamide by assessing the occurrence of dose limiting toxicities | 12 months

SECONDARY OUTCOMES:
Measurement of plasma levels of study drug to determine the pharmacokinetic properties of MM-398 in combination with cyclophosphamide | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Harker-Murray, MD, Study Chair — Midwest Children's Hospital
Locations (6):
- United States (6):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - UT Southwestern, Dallas, Texas
  - MD Anderson Children's Cancer Hospital, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Midwest Children's Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903